CLINICAL TRIAL: NCT03921203
Title: ApoB48IC2 Metabolism in Plasma and Interstitial Fluid
Brief Title: ApoB48 Metabolism in Plasma and Interstitial Fluid
Status: Completed | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Responsible Party: Principal Investigator, Mats Rudling, Professor, Karolinska University Hospital
Other Study IDs: ApoB48IC2
Record Dates: First submitted 2019-04-17; First posted 2019-04-19 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Interstitial fluid and blood (serum, plasma and whole blood)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Type 2 diabetes patients
- Healthy controls

SUMMARY:
Postprandial increases in the levels of atherogenic chylomicron remnant lipoprotein particles have long been considered a presumable risk factor for the development of atherosclerosis with time, also in normolipidemic subjects. apoB-48 (Chylomicron) in blood is a specific marker for intestinal derived lipoproteins. Specific aim: To determine if apoB-48 containing lipoproteins may appear in IC in the postprandial state after a standard meal and investigate the effect fasting and feeding have on levels of lipids, apolipoproteins and the cholesterol component of lipoproteins in IF and plasma.

Methodology: Intercellular fluid will be collected using the cup technique. IF will be collected in intervals corresponding to different periods after food intake. The IF from these different occasions will then be analysed and compared using FPLC and Elisa.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years.
* For the T2D study group: Diagnosed with type 2 diabetes.

Exclusion Criteria:

For subjects with type 2 diabetes:

* Systemic inflammatory disease that requires active treatment
* Thyroid disease that requires active treatment
* Skin disease that requires active treatment and causes significant changes in the area of the skin that is to be investigated
* Treatment with oral glucocorticoids
* Levels of SR, TSH, T4 or Hemoglobin in the blood pronouncedly outside the reference range
* Pregnancy

For healthy controls:

* Registered disease in the health declaration that requires continuous systemic treatment. Exception to the above: well controlled hypertension in which case the subject should not have treatment with more than one antihypertensive drug, the drug must not be an alpha-blocker or beta-blocker or thiazide diuretic
* Skin disease that requires active treatment and causes significant changes in the area of the skin that is to be investigated
* Blood pressure pronouncedly above 140/90
* Blood test results pronouncedly outside the reference range
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy controls and type 2 diabetes patients over 18 years old, matched for age and gender.
Sampling Method: Non-Probability Sample
Enrollment: 22 (Actual)
Dates: Start 2019-04-17 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
ApoB48 levels in blood and interstitial fluid | 7 hours

CONTACTS AND LOCATIONS:
Overall Officials: Mats Rudling, Principal Investigator — Karolinska Institutet
Locations (1):
- Patient research centre, Clinic of endocrinology, Karolinska University Hospital, Stockholm, Huddinge, Sweden